CLINICAL TRIAL: NCT05497193
Title: Clinical Efficacy and Safety of Perampanel Monotherapy in the Treatment of Children With Focal Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yang Xinwei (Other)
Responsible Party: Sponsor-Investigator, Yang Xinwei, Deputy Chief Physician, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: 20222126
Record Dates: First submitted 2022-07-26; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — perampanel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: perampanel — China's state food and drug administration approved indications for adults and children aged 4 or more focal epileptic hair company or not with secondary comprehensive seizures of epilepsy, adding treatment, in July 2020 to monotherapy without clinical approval, the current domestic perampanel monotherapy clinical effectiveness and safety of focal epilepsy in children have not been reported.
  Other Names: No other interventions currently

SUMMARY:
This project is a multicenter prospective study. By retrieving outpatient medical records and collecting clinical data of epilepsy patients, the efficacy and safety of single-drug perampanel in patients with focal epilepsy were analyzed.

DETAILED DESCRIPTION:
This project is a multicenter prospective study. The selected case population was given the oral antiepileptic drug perampanel for 12 months, and the seizure control (complete control, markedly effective, effective, ineffective, worsening), EEG changes (normal, Effective, ineffective), and adverse reactions were analyzed, so as to provide a basis for perampanel monotherapy in children with focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

(1) Clinical diagnosis of focal epilepsy; (2) Take anti-epileptic drugs as prescribed by your doctor; (3) Epilepsy patients diagnosed with focal epilepsy with or without generalized seizures, and Monitoring for ≥12 months; (4) Newly diagnosed epilepsy patients, or only taking 1-2 other AEDs, without regular antiepileptic treatment, the efficacy is not good, after using perampanel, gradually stop AEDs for 8 weeks. For perampanel monotherapy; (5) the number of seizures ≥ 1 in the first 3 months of enrollment.

Exclusion Criteria:

(1) syncope (2) Pseudo-seizure(3)transient ischemic attack

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients in the pediatric outpatient department of our hospital
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy after drug treatment: | one year
  Epilepsy seizures: the seizure frequency 3 months before treatment is the baseline, and the maintenance period is compared with the baseline. Complete control: no seizures after treatment; markedly effective: seizure frequency reduced by > 75%; effective: seizure frequency reduced by > 51%-74 %; Ineffective: frequency reduced by ≤50%, worsening: attack frequency increased by 25%.
EEG changes after drug treatment | one year
  EEG changes: (1) normal EEG (2) abnormal EEG: including epileptiform discharge, background rhythm slowing, epileptiform discharge + background rhythm slowing. EEG judgment: (1) normal: the epileptiform discharge disappeared or the background slowing disappeared (2) effective: the epileptiform discharge was reduced or the background slowing was improved (3) invalid: the epileptiform discharge did not change or aggravate after the drug.
safety after drug treatment | one year
  Common adverse reactions include: dizziness, drowsiness, fatigue, irritability, nausea and falls and weight gain.

CONTACTS AND LOCATIONS:
Overall Officials: xinwei yang, doctor, Principal Investigator — hospital doctor
Locations (1):
- XI Jing Hospital, Xi'an, Shaanxi, China